CLINICAL TRIAL: NCT02767245
Title: Efficacy of Thiamine Supplement for Improve Cardiovascular Function in Patients With Severe Hyperthyroidism
Brief Title: Thiamine Supplement in Patients With Severe Hyperthyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Chutintorn Sriphrapradang, Assistant Professor, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-56-10
Record Dates: First submitted 2016-05-09; First posted 2016-05-10 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Thyrotoxicosis
Keywords: Thiamine; Congestive heart failure; Atrial fibrillation; Graves' disease
MeSH Terms: conditions — Thyrotoxicosis; Heart Failure; Atrial Fibrillation; Graves Disease | interventions — Thiamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thiamine (Active Comparator): Thiamine intravenously 100 mg/day for 3 days
  Interventions: Drug: Thiamine
- No thiamine (No Intervention): No thiamine was given to the patient

INTERVENTIONS:
Drug: Thiamine — Thiamine IV 100 mg/day
  Other Names: vitamin B1
  Arms: Thiamine

SUMMARY:
Thyrotoxicosis is a hypermetabolic state in which there is increased utilization of thiamine. Thiamine deficiency has been observed in association with hyperthyroidism. Several studies documented that thiamine treatment could improve signs and symptoms of congestive heart failure, or even improve left ventricular ejection fraction in patients without thyrotoxicosis. This pilot study aims to evaluate prevalence of thiamine deficiency and assess improvement of cardiovascular function after receiving thiamine supplement in thyrotoxic patients.

DETAILED DESCRIPTION:
The prevalence of thiamine or vitamin B1 deficiency has been documented in 21-98% of patients with heart failure. Thiamine has multiple effects on the cardiovascular system. It has important hemodynamic effects on the circulatory system as well as direct positive pharmacologic effects on the heart. Thiamine deficiency has been shown to cause cardiac hypertrophy, depressed cardiac contractility, and dysrhythmias. Thiamine is of particular interest in the management of heart failure for several reasons. Heart failure is a disease of the elderly whose micronutrient status is in need of attention. Heart failure patients tend to have inadequate nutrient intake, which has been associated with thiamine deficiency. Use of loop diuretic is associated with the loss of water-soluble vitamins, including thiamine. Several studies have examined the role of thiamine supplementation in patients with heart failure. Clinical trials in patients with congestive heart failure have shown that thiamine supplementation increases the systolic, diastolic, and central venous pressures, with a decline in heart rate and increase in left ventricular ejection fraction (LVEF). Thiamine acts as a vasodilator and reduces the afterload on the heart, thus improving cardiac function. Thiamine has also been reported to increase diuresis and natriuresis in patients with heart failure receiving diuretics.

Thyrotoxicosis considerably increases the demand for thiamine. In vivo study in a rat model demonstrated that thyroid hormones have a direct influence on mitochondria which is the main source of energy. Thiamine in its various forms functions as an important coenzyme for macronutrient oxidation and the production of adenosine triphosphate. Thiamine pyrophosphate works in several oxidative decarboxylation reactions and is a catalyst in the reactions of Krebs cycle. Therefore, thiamine seems to decrease in the case of an increased tissue metabolism. In the previous case reports, they described the possible association between thyrotoxicosis and thiamine deficiency in patients manifested as Wernicke-Korsakoff syndrome.

Despite lack of the evidence of benefit of thiamine therapy in patients with severe thyrotoxicosis or thyroid storm, some experts recommended thiamine in conjunction with other supportive treatment. We aimed to investigate the effect of thiamine on cardiac function in patients with severe thyrotoxicosis in a prospective, randomized, open, blinded end-point study using echocardiographic as well as clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with severe thyrotoxicosis
* Thyrotoxic patients with cardiovascular involvement e.g. heart rate > 90/min, atrial fibrillation or congestive heart failure
* Agree to participate by written informed consent

Exclusion Criteria:

* Previously treated with thiamine within 1 month before the enrollment
* End-stage renal disease
* Alcoholism
* Pregnant or lactating women
* Post gastric bypass surgery

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
left ventricular systolic function | 3 months
  Left ventricular systolic function was assessed by using transthoracic 2-dimension echocardiography. The measurement was followed the standard protocol of American Society of Echocardiography including wall thickness, left ventricular size and mass and left ventricular ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Chutintorn Sriphrapradang, M.D., Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided